CLINICAL TRIAL: NCT04004962
Title: Use of Infrared Spectroscopy in Fast Septic Arthritis Diagnosis
Acronym: SYNOFRESH
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_8857_SYNOFRESH
Record Dates: First submitted 2019-06-25; First posted 2019-07-02 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-03

CONDITIONS: Joint Effusion
MeSH Terms: conditions — Hydrarthrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Infrared spectroscopy — Infrared spectroscopy

SUMMARY:
To study the diagnostic performance of infrared spectroscopy on fresh synovial fluids in early septic arthritis diagnosis in patients with acute joint effusion

DETAILED DESCRIPTION:
Diagnosis of a joint effusion is frequently a medical emergency, especially when septic arthritis is suspected. Septic arthritis diagnosis relies on microscopic and bacteriological analysis of synovial fluid obtained by arthrocentesis. Direct microscopic examination can be made within 2 to 12 hours but it is negative in about 50 % of the cases. It is necessary to wait 72 hours to obtain the result of the culture and reasonably rule out the diagnosis of septic arthritis. A method of establishing an immediate etiological diagnosis could improve the care of patients with joint effusion that is a therapeutic emergency and justify a hospitalization and a parenteral antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 year old
* patients with an acute arthritis defined by an evolution of less than 6 weeks
* patients benefiting from joint fluid puncture for diagnostic purposes in the rheumatology hospitals participating in the study
* patients who received information about the protocol and have not expressed opposition to participate

Exclusion Criteria:

* patients opposing the study
* protected major (safeguard justice, trusteeship and guardianship) and persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients benefiting from joint fluid puncture for diagnostic purposes in the rheumatology hospitals participating in the study
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Diagnosis of the cause of joint effusion | Up to 7 days (time to perform Spectroscopy and collect laboratory results)
  The final diagnosis of the cause of joint effusion is made by the clinician based on the clinical and laboratory data : septic arthritis or other causes of arthritis

SECONDARY OUTCOMES:
Number of days of hospitalization | Up to 2 months (time to collect data on hospitalization duration and antibiotic therapy duration)
  The clinician will be asked to state how a positive or a negative result of the diagnostic test under study would have affected his decision to hospitalize the patient
Total dose of antibiotics | Up to 2 months (time to collect data on hospitalization duration and antibiotic therapy duration)
  The clinician will be asked to state how a positive or a negative result of the diagnostic test under study would have affected his decision to start antibiotic therapy

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Angers, Angers
  - CHRU Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Nantes, Nantes
  - CHU de Rennes, Rennes
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No